CLINICAL TRIAL: NCT02470962
Title: Cardiac Involvement in Patients With Duchenne/Becker Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: DMD-Herz
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Duchenne / Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with muscular dystrophy: Boys aged 8 to 18 years with muscular dystrophy of the Duchenne / Becker type
- Children without heart disease: Children without heart disease, aged 8-18 years, as CMR comparison group
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation by serial echocardiography with extended techniques and cardiac magnetic resonance imaging
  Groups: Children without heart disease

SUMMARY:
This study evaluates the function of the heart in young patients with muscular dystrophy type Duchenne or Becker. Participants have their hearts examined at regular intervals by ultrasound (echocardiography) and cardiac magnetic resonance imaging.

DETAILED DESCRIPTION:
Muscular dystrophy leads to progressive loss of function in all muscles during childhood and adolescence, including the heart. The usual method to evaluate the heart is echocardiography, emphasizing few parameters. Cardiac magnetic resonance imaging is not as widely available as echocardiography, but early changes can be detected before they become visible on echocardiography. In this study, the investigators compare the methods of measuring heart function in order to find the best measurements for follow up and to see how fast the degenerative changes occur in the hearts of patients with muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged 8 to 18 years with DMD/BMD confirmed genetically or by muscle biopsy
* Informed consent

Exclusion Criteria:

* Other clinically significant concomitant disease states (e.g., renal failure)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant or his/her parents or legal caregivers,
* Inability to lie still for the duration of the imaging procedures (approximately 45 minutes each for echocardiography and CMR)
* MR-incompatible implanted or accidentally incorporated metal device or claustrophobia that prohibits use of magnetic resonance imaging

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Boys aged 8 to 18 years with DMD/BMD confirmed genetically or by muscle biopsy
  * Control group for CMR: children without heart disease
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 3 years per patient

SECONDARY OUTCOMES:
Quantification of fibrosis by LGE/T1 mapping | 3 years per patient
NT-proBNP | 3 years per patient

CONTACTS AND LOCATIONS:
Overall Officials: Barbara EU Burkhardt, MD, Principal Investigator — Children's Hospital Zürich, Switzerland
Locations (1):
- Children's Hospital, Zurich, Canton of Zurich, Switzerland